CLINICAL TRIAL: NCT04405531
Title: Effectiveness of Task-Oriented Training on Occupational Performance, Independence, and Fatigue in Children With Childhood Cancer: A Randomized-Controlled Trial
Brief Title: Effects of TOT on Performance, Independence and Fatigue in Children With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ZEYNEP KOLİT, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KCTOT
Record Dates: First submitted 2020-05-16; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Childhood Cancer; Performance; Functional Independence; Fatigue
Keywords: childhood cancer; fatigue; functional independence; occupational performance; task-oriented training
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- task-oriented training(TOT) (Experimental): The first phase of the TOT, functional activity analysis, was performed for the activities, for which performance problem was determined by Canadian Occupational Performance Measure (COPM) and Functional Independence Measure for Children (WeeFIM). In the second phase, the occupational performance, fatigue and functional independence levels that prevent the realization of the activity were determined by functional activity analysis. These designated occupational performance, fatigue and functional independence levels constitute the task of this study, as we aim to improve children's functionality. In the third phase, various functional activities including these tasks were executed. The TOT was practiced by following the above mentioned steps for each performance area. All the activities were designed for the inpatient settings of children.
  Interventions: Other: task-oriented training (TOT); Other: conventional occupational therapy (COT)
- conventional occupational therapy (COT) (Experimental): The treatment efficacy determined by the therapist was provided by considering the functional level in order to achieve the desired goal by the participant. The COT included functional activities based on the client-centered principles of the neuro-developmental approach. All the sessions started with relaxation training combined with breathing exercises. At the end of approximately 10 minutes of application time, individualized functional activities were implemented.
  Interventions: Other: conventional occupational therapy (COT)

INTERVENTIONS:
Other: task-oriented training (TOT) — The study group received a TOT together with a conventional occupational therapy (COT). The study groups received a treatment for 20 sessions at a hospital setting.
  Other Names: TOT
  Arms: task-oriented training(TOT)
Other: conventional occupational therapy (COT) — The control group received only a COT program. The control groups received a treatment for 20 sessions at a hospital setting.
  Other Names: COT

SUMMARY:
This study aims to explore the effects of Task-Oriented Training (TOT) on occupational performance, activities of daily living and fatigue of children in pediatric oncology clinic.

Hypothesis: There is no effect of TOT on occupational performance and satisfaction in children with childhood cancer. There is no effect of TOT on functional independence in daily living activities in children with childhood cancer. There is no effect of TOT on fatigue levels in children with childhood cancer.

ELIGIBILITY:
Inclusion Criteria:

* being between 6 and 14 years of age;
* receiving inpatient chemotherapy sessions;
* having taken scores higher than 28, 30 and 35 in the mini-mental state exam devised for children of ages 6-8, 9-11 and 12-14, respectively.

Exclusion Criteria:

* their disease had recurred, or they were in palliative care;
* they or their parents were not fluent speakers of the Turkish language;
* they were unwilling to take part in the programs.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 213 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 6 months
  COPM is a standard measurement used for measuring the occupational performance and satisfaction in children by identifying their problems in performing activities of daily living. Each of the identified activities was asked to be scored between 1 and 10 on the Likert Scale (1: not important; 10: very important). Performance and satisfaction scores were specified by dividing the total scores of performance and satisfaction to the number of activities that the children regard as substantial. A change of two points or more in the score on COPM is considered clinically significant. In the Turkish version of validity and reliability, the internal consistency coefficient of COPM was found to be between 0.9 and 1.
Functional Independence Measure for Children (WeeFIM) | 6 months
  WeeFIM, which is an 18-item and seven-level ordinal scale, measures a child's incoherent performance in basic daily functional skills. It can be used for children with developmental disabilities from 6 months to 21 years. Sub-scales include self-care, sphincter control, movement, transfers, social cognition and communication. The self-care subscale has six items: eating, grooming, bathing, dressing of upper and lower extremities, and the perineal hygiene and adjustment of necessary clothes for the toilet. A scoring scale between 1 (total assistance) to 7 (total independence) was used at this steep. The maximum total score is 126 and the lowest total score is 18, while the maximum scores for self-care, mobility, and cognition are 56, 35, and 35, respectively .
Visual analog scale (VAS) | 6 months
  VAS is a reliable and easily applicable assessment tool that is accepted worldwide in the literature. VAS is used to transform some immeasurable values into quantitative data. It is a scale in which a person marks his / her current emotion level on a vertical line with a 10-cm scale. Every emotion is evaluated in a range from non-existent (i.e. never experiencing that particular sensation or feeling) to highly intensive (i.e. constantly experiencing that particular sensation or feeling). The following expressions were used on the scale: 'Show me your fatigue level on the line, here is no fatigue (score = 0), and there is the wickedest probable fatigue (score = 10)'. This process was repeated for five times as before activity, during-activity, after activity, and morning and evening time intervals. It took less than 1 minute for each application to get completed.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Kolit, MSc, Principal Investigator — Hacettepe University; Sedef Şahin, PhD, Study Director — Hacettepe University; Ceren Davutoğlu, MSc, Principal Investigator — Hacettepe University; Meral Huri, PhD, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No